CLINICAL TRIAL: NCT03544359
Title: Longitudinal Functional MRI Study of Transcranial Electrical Stimulation in Chronic Tinnitus
Brief Title: MRI Study of Noninvasive Transcranial Electrical Stimulation in Tinnitus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Amber Leaver, Research Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00207056; R21DC015880 (NIH)
Record Dates: First submitted 2018-05-07; First posted 2018-06-01 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Tinnitus, Subjective
Keywords: transcranial direct current stimulation (tDCS); functional magnetic resonance imaging (MRI)
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Eligible volunteers will be randomly assigned to receive either 5 consecutive days of active tES or 5 consecutive days of sham/inactive tES. This part of the study is optional. All eligible volunteers will receive active and sham/inactive tES during MRI.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tES (Active Comparator)
  Interventions: Device: Transcranial electrical stimulation (tES)
- Sham/Inactive tES (Sham Comparator)
  Interventions: Device: Transcranial electrical stimulation (tES)

INTERVENTIONS:
Device: Transcranial electrical stimulation (tES) — In tES, a mild electrical current is passed between two or more electrodes placed on the volunteer's head (scalp). In this study, a mild unvarying (constant) electrical 2mA current is passed between two rubber electrodes placed on the head over auditory cortex for 20 minutes per session for 5 consecutive days. Because the electrical current direction (positive/negative) and current amplitude (2mA) does not vary or change during stimulation, this type of tES is also called transcranial "direct current" stimulation, or tDCS.
  Other Names: Transcranial direct current stimulation (tDCS)

SUMMARY:
The purpose of this research is to understand how a neuromodulation technique, transcranial electrical stimulation (tES), affects brain function in adults with chronic tinnitus measured with functional magnetic resonance imaging (fMRI). We hypothesize that multiple sessions of tES (5 consecutive days) will modulate:

1. Overall activity and local connectivity within brain regions near tES electrodes, and
2. Functional connectivity within brain networks associated with brain regions near tES electrodes.

In exploratory analyses, we also measure the extent to which the hypothesized changes listed above a related to changes in tinnitus symptoms after tES.

DETAILED DESCRIPTION:
Chronic subjective tinnitus is a common and sometimes disabling condition, with few effective treatments and no cure. Tinnitus is thought to involve dysfunction in central brain networks subsequent to peripheral injury or interference; thus, neurostimulation therapies that directly target central circuits are receiving growing interest. Of these, noninvasive transcranial electrical stimulation (tES) is an attractive option, due to its relative affordability, mobility, and favorable safety profile. A growing number of studies have demonstrated that tES of temporal/auditory cortex is effective at transiently reducing tinnitus symptoms, including tinnitus loudness and tinnitus distress. However, the results of previous clinical trials are variable, and a mechanistic understanding of tES and its therapeutic effects remains elusive. The main goal of this research is to lay the groundwork for improved, patient-centered approaches to noninvasive neurostimulation therapy for chronic tinnitus. To accomplish this long-term goal, this study will determine how the intrinsic activity and connectivity of auditory networks are affected during simultaneous tES-fMRI of auditory cortex, specifically in those patients who experience reduced tinnitus symptoms after 5 consecutive days of tES. Though the primary goal of the proposed research is to optimize tES for the treatment of tinnitus, these studies will also provide a wealth of information regarding tinnitus pathophysiology and the mechanisms of tES more generally, which is being investigated for the treatment of a wide variety of brain disorders and injuries.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 65
* Race/ethnicity: all races and ethnic groups
* Sex/Gender: all
* Capacity to provide informed consent
* Subjective tinnitus symptoms for at least one year prior (confirmed by patient self-report)
* Has discussed tinnitus symptoms with clinician (i.e., physician, audiologist) to confirm low/no likelihood of physical or neurological origin of tinnitus symptoms (e.g., acoustic neuroma, Meniere's Disease, etc.), confirmed by patient self-report
* Stable standard or no pharmacological treatment regimen for tinnitus (e.g., SSRI or SNRI) with no change in treatment 6 weeks prior to study start

Exclusion Criteria:

* Ages below 18 (neurobiology is quite different in children vs. adults)
* Ages above 65 (cortical excitability changes with age)
* Tinnitus symptoms with known medial origin, including: Meniere's disease, pulsatile tinnitus, acoustic neuroma, spontaneous optoacoustic emissions, any other known medical origin
* Diagnosis of any medical condition potentially affecting brain function, including: neuropsychiatric or mental disorders, mood disorders (bipolar disorder, anxiety, PTSD), psychotic states or disorders, developmental disorders, neurological disorders, including mild cognitive impairment, significant head injury, significant history of alcohol/substance abuse or dependence, chronic pain (>1 year duration)
* MRI contraindications: metal or other implants that are not MR-safe, claustrophobia, pregnancy or suspected pregnancy
* tDCS contraindications*: skin conditions or injuries on the scalp, hair extensions, wigs, braids, etc. that cannot be removed prior to the study, metal implants or pacemakers (also contraindicated for MRI) *Please note that history of seizures or epilepsy, stroke, and brain injury are not safety concerns for tES use, and may be inclusion criteria for other tES studies. However, individuals with history of these conditions will be excluded here because these conditions are not a focus of the current study (see above).
* Non-English speakers (due to written consent and questionnaires administered)
* other major medical conditions (e.g., cancer, stroke).
* Significant history of alcohol/substance abuse or dependence within last 12 months
* Neurostimulation or neuromodulation treatment for any reason within the past 3 months
* Current medication use potentially affecting brain function, including decongestants, antihistamines, benzodiazepines or other anticonvulsants, anti-psychotics, or antidepressants.
* Prisoners will not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Changes in brain function (functional connectivity) | baseline, interim (1 week after baseline), and post-tES (2 weeks after tES)
  Changes in temporal coherence (functional connectivity) of local auditory-cortex activity and auditory networks measured with BOLD-fMRI

SECONDARY OUTCOMES:
Tinnitus loudness ratings | daily from date of randomization until 2 weeks after the the last study visit (tES session)
  Perceived loudness of tinnitus sensation will be measured using a 10-point Likert rating scale, where a rating of "1" indicates no tinnitus and a rating of "10" indicates loudest tinnitus imaginable. In this rating scale, higher ratings indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Translational Imaging, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified research data may be shared upon completion of the study with researchers according to Northwestern IRB approved protocols. Shared data will not include personally identifiable information or protected health information.
Time Frame: After study completion, data will be made available upon request and upon approvals from all relevant regulatory agencies.
Access Criteria: Approval of Institutional Review Board (and/or other relevant regulatory agencies) at all involved institutions.